CLINICAL TRIAL: NCT00209131
Title: Efficacy of Flomax to Improve Stone Passage Following Shock Wave Lithotripsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to frequent turnover of research coordinators and thus poor study accrual.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kenneth Ogan, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0128-2005
Record Dates: First submitted 2005-09-14; First posted 2005-09-21 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-09

CONDITIONS: Urolithiasis
Keywords: urolithiasis
MeSH Terms: conditions — Urolithiasis | interventions — Tamsulosin; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flomax (Experimental): Patients on this arm will be given 0.4mg of Flomax to be taken for one month following their shock wave lithotripsy procedure.
  Interventions: Drug: Flomax
- Sugar pill (Placebo Comparator): Patients on this arm will be given a sugar pill to be taken for one month following their shock wave lithotripsy procedure.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Flomax — 0.4mg Flomax pills will be given to patients to take once daily for one month following shock wave lithotripsy to aid the stone passage.
  Other Names: Tamsulosin
  Arms: Flomax
Drug: Sugar pill — Comparable sugar pills will be given to the placebo group to take daily for one month following shock wave lithotripsy to aid stone passage.
  Other Names: Placebo pill
  Arms: Sugar pill

SUMMARY:
The majority of kidney stones are treated with shock wave lithotripsy (SWL). We are examining if the medication Flomax will result in improved stone passage rates following SWL.

DETAILED DESCRIPTION:
Placebo blinded study examining the effects of Flomax on stone passage rates following SWL.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and above with urolithiasis scheduled for shock wave lithotripsy.

Exclusion Criteria:

* Contraindications to Flomax
* Patients with renal impairment (serum creatinine above 2.0)
* Patients with hepatic impairment (liver enzymes 2.5 times the upper limit of normal)
* Use of other oral alpha blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Ogan, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment took place in a medical clinic affiliated with a teaching hospital from May 2005 through February 2009.
Period: Overall Study
Arm/Group | Flomax | Sugar Pill
Started | 15 (Patients enrolled for participation but did not complete the study.) | 11 (Patients enrolled for participation but did not complete the study.)
Completed | 0 (Lack of personnel for adequate followup and data collection.) | 0 (Lack of personnel for adequate followup and data collection.)
Not Completed | 15 | 11
Not completed — Lack of personnel due to turnovers. | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flomax | Sugar Pill | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 11 | 26
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55 (5) | 53 (5) | 54 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Passage of Stone Fragments
Description: Time to passage of stone fragments following shock wave lithotripsy as documented by patient diaries and follow-up radiographic imaging.
Time Frame: 2 weeks and 3 months
Population: No analysis was conducted.
Arm/Group | Flomax | Sugar Pill
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Flomax vs Sugar Pill; No analysis was conducted; Test type: Non-Inferiority or Equivalence; p < 0.05, Other

2. Secondary Outcome: Medical Evaluation
Description: Evaluation of pain assessments, lower urinary tract symptoms, side effects of study medication and need for hospitalizations and additional endoscopic procedures.
Time Frame: 2 weeks and 3 months
Arm/Group | Flomax | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Flomax | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study was terminated due to turnovers of personnel to assist with recruitment and execution of the study.Recruitment was strained and patients recruited could not be followed up in a timely fashion to adhere to protocol. Thus, no data was generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No